CLINICAL TRIAL: NCT05602493
Title: A Randomized Control Trial Phase (IIIa) Unicentric, Placebo Controlled, Double-Blinded Study to Confirm the Efficacy and Safety of 'Topical Alendronic Acid on Alveolar Bone Remodeling After Tooth Extraction: a Pilot Study´
Brief Title: A Randomized Control Trial Phase (IIIa) Unicentric, Placebo Controlled, Double-Blinded Efficacy and Safety of Topical Alendronic Acid on Alveolar Bone Remodeling After Tooth Extraction
Acronym: XEOLAS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xeolas Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XeolasPharma
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bone Loss, Alveolar
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Clinical Trial Phase (IIIa), Unicentric, Placebo Controlled, Double-Blinded Study"
Who Masked: Participant, Investigator
Masking Description: Double-Blinded Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (n=30) Soludronate® 0.7 mg/ml (Experimental): It will be applied on the fresh extraction socket for 15 min and then rinsed with sterile saline 3 time, 1 minute each rinse. After the extraction will be required a CBCT scan. The medication that will be prescribed for the patient will be Enantyum 25 mg (2-3 days) and in case of allergic patient Paracetamol 650 mg (2-3 days).
  15 days later (-/+ 2 days), during the follow-up 1 the suture will be removed, the cicatrization of the surgical site evaluated and intraoral photos will be taken. The last follow-up (2) visit, 91 days later (-/+ 2 day) the follow-up 2 will take place. A CBCT scan and intraoral photos will be required.
  Interventions: Drug: Soludronate®
- control group (n=30) sterile saline (Placebo Comparator): It will be applied on the fresh extraction socket for 15 min and then rinsed with sterile saline 3 time, 1 minute each rinse. After the extraction will be required a CBCT scan. The medication that will be prescribed for the patient will be Enantyum 25 mg (2-3 days) and in case of allergic patient Paracetamol 650 mg (2-3 days).
  15 days later (-/+ 2 days), during the follow-up 1 the suture will be removed, the cicatrization of the surgical site evaluated and intraoral photos will be taken. The last follow-up (2) visit will be 1,5 months after the intervention and will be optional for those cases showing redness, swelling or pain during the first follow up, 3,5 months later (-/+ 1 week) the end visit will take place. A CBCT scan and intraoral photos will be required at the end visit.
  Interventions: Drug: sterile saline

INTERVENTIONS:
Drug: Soludronate® — In the first visit, the randomized process will take place. Tooth extraction procedure will be performed.
  Arms: test group (n=30) Soludronate® 0.7 mg/ml
Drug: sterile saline — sterile saline
  Arms: control group (n=30) sterile saline

SUMMARY:
The purpose of the study is to determine the efficacy and safety of the effects of a topical medication on bone remodeling after dental extraction, in order to establish whether such treatment can be a new therapeutic option for said pathology. The participation of 60 patients is expected, who will be divided randomly in equal proportions into two groups. Treatment groups: Group A (30 patients): medication administered topically. Group B (30 patients): placebo with characteristics equal to the drug under investigation.

DETAILED DESCRIPTION:
The purpose of the study is to determine the efficacy and safety of the effects of a topical medication on bone remodeling after dental extraction, in order to establish whether such treatment can be a new therapeutic option for said pathology. The participation of 60 patients is expected, who will be divided randomly in equal proportions into two groups. Treatment groups: Group A (30 patients): medication administered topically. Group B (30 patients): placebo with characteristics equal to the drug under investigation. Subsequently, a review will be carried out 15 days later to assess the status of the intervention performed and a final visit 3 months after surgery. Neither the doctor nor the patient will know what treatment they will receive during the study. You will have a 50% chance of receiving the placebo, which will have the same characteristics in terms of color, texture and consistency; but it does not contain the pharmacologically active substance and therefore it is not expected to have an effect. Before the start of the study, it will be assessed if you accomplish the criteria of the study, you will be informed of all doubts and you must sign the patient informed consent form. You will need to attend study visits: Your participation in the study will last approximately 3.5 months. Throughout which you will have to go four times to the University Dental Clinic. On the 1st visit, the treatment group will be assigned together with dental extraction and application of the medication or placebo for 15 min. and you will have to rinse 3 times for 1 min. with sterile saline solution. A cone beam computed tomography (CBCT) scan will be performed and photos will be taken. The 2nd visit will take place after 15 days where the suture stitches will be removed and a review will be carried out where photos will be taken to assess the evolution. At approximately 3.5 months, both the imaging test (CBCT) and the photos will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form.
* Overall, healthy patients that qualify for oral surgery (ASA I and II).
* Male and female patients 18-90 (inclusive) years of age.
* Requiring extraction of 1 tooth (maxillary or mandibular).
* Stable post-extraction socket walls with at least 4 walls.
* Adequate oral hygiene: plaque index < 25% before the surgery.
* Non-smoker or smoker of <10 cigarettes per day.
* Able to follow the instructions and able to meet the follow-ups.
* Healthy or controlled periodontal disease.

Exclusion Criteria:

* Patients who do not agree with informed consent.
* Male and female patients are not 18-90 (inclusive) years of age. Patients taking medication that can interfere with the treatment such as Calcium Carbonate or Vitamin D.
* Untreated periodontal disease.
* Presence of dehiscence and/or fenestration at buccal plate of the extraction tooth/teeth.
* Patient who will need guided bone regeneration (GBR) or Block Regeneration after the extraction.
* History of head and/or neck radiation.
* History of chemotherapy in the five years prior of the surgery.
* Non controlled Diabetes.
* Chronic corticoids medication that may influence healing and/or osseointegration.
* Smoker of >10 cigars per day.
* Pregnant woman
* Alcohol or drugs.
* Patient going under bisphosphonates treatment or taking Denosumab (Prolia®).
* Patient with diagnosed osteoporosis, hypocalcemia, hypersensibility to alendronic acid or any of the excipients of Soludronate®.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Buccal and lingual vertical and horizontal bone socket dimensions will be measured by CBCT. | Day 1
  Three dimensional volumetric changes in hard tissue will be measured in (mm).

SECONDARY OUTCOMES:
Record any adverse effect and their severity related to the Soludronate® or its use. | 1 day to 3 months
  First follow-up: assessments to be performed during the visit: control, suture removal, photos and evaluation of the surgical site at 15 days.
  Second follow-up: optional visit, 1,5 months after the treatment. If the patient shows abnormal redness, swelling or pain in the first follow up, patient will be scheduled for a second visit.
  End of the study: assessments to be performed during the visit: CBCT scan and intraoral photos at 3,5 months approximately after the treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis McDaid, PhD, Study Director — Xeolas Pharmaceuticals Ltd
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain